CLINICAL TRIAL: NCT03400839
Title: Investigation of the Impact of Clinical Outcomes on Disease Progression and Prognosis in Patients With Interstitial Lung Diseases
Brief Title: Best Clinical Endpoints That Likely Induce Worse Prognosis in Interstitial Lung Diseases
Acronym: BELIEVE-ILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: Universidade Norte do Paraná (Other)
Responsible Party: Sponsor
Other Study IDs: 2.143.496
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-11

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial Lung disease; prognosis; clinical endpoints; association
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Walk Test; Exercise Test; Respiration; Body Composition; Oxidative Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Clinical and biological data collected in the study may be used in other investigations upon participants written consent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ILD: Patients with a medical diagnosis of interstitial lung disease.
  Patients will be submitted to the assessment of:
  * Daily physical activity levels;
  * 6-minute walk test;
  * Cardiopulmonary exercise testing;
  * Muscle Function;
  * Lung Function;
  * Body composition;
  * HRQoL - SGRQ-I;
  * HRQoL - SF36;
  * Anxiety and depression;
  * Symptoms - mMRC
  * Symptoms - UCSD/SOBQ;
  * Sleep quality;
  * Sleepiness;
  * Inflammatory markers and oxidative stress.
  * Functional performance tests
  Interventions: Diagnostic Test: Daily physical activity levels; Diagnostic Test: 6-minute walk test; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Muscle Function; Diagnostic Test: Lung Function; Diagnostic Test: Body composition; Diagnostic Test: HRQoL - SGRQ-I; Diagnostic Test: Symptoms - UCSD/SOBQ; Diagnostic Test: HRQoL - SF36; Diagnostic Test: Anxiety and depression; Diagnostic Test: Symptoms - mMRC; Diagnostic Test: Sleep quality; Diagnostic Test: Sleepiness; Diagnostic Test: Inflammatory markers and oxidative stress; Diagnostic Test: Functional performance tests
- Control Group: Age-matched peers without lung diseases.
  Participants will be submitted to the assessment of:
  * Daily physical activity levels;
  * 6-minute walk test;
  * Cardiopulmonary exercise testing;
  * Muscle Function;
  * Lung Function;
  * Body composition;
  * HRQoL - SF36;
  * Anxiety and depression;
  * Sleep quality;
  * Sleepiness;
  * Inflammatory markers and oxidative stress.
  * Functional performance tests
  Interventions: Diagnostic Test: Daily physical activity levels; Diagnostic Test: 6-minute walk test; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Muscle Function; Diagnostic Test: Lung Function; Diagnostic Test: Body composition; Diagnostic Test: HRQoL - SF36; Diagnostic Test: Anxiety and depression; Diagnostic Test: Sleep quality; Diagnostic Test: Sleepiness; Diagnostic Test: Inflammatory markers and oxidative stress; Diagnostic Test: Functional performance tests

INTERVENTIONS:
Diagnostic Test: Daily physical activity levels — Objectively measured physical activity using activity monitors.
Diagnostic Test: 6-minute walk test — Assessment of functional exercise capacity.
Diagnostic Test: Cardiopulmonary exercise testing — Assessment of maximal exercise capacity.
Diagnostic Test: Muscle Function — Assessment of muscle force, muscle endurance and muscle fatigability
Diagnostic Test: Lung Function — Assessment of whole-body plethysmography and spirometry.
Diagnostic Test: Body composition — Assessment of bioelectrical impedance.
Diagnostic Test: HRQoL - SGRQ-I — Assessment of Health-related quality of life by the "Saint-George Respiratory questionnaire (SGRQ-I)"
  Groups: Patients with ILD
Diagnostic Test: Symptoms - UCSD/SOBQ — Assessment of symptoms by the "UCSD Short of breath questionnaire"
  Groups: Patients with ILD
Diagnostic Test: HRQoL - SF36 — Assessment of Health-related quality of life by the "SF-36 questionnaire"
Diagnostic Test: Anxiety and depression — Assessment of anxiety and depression by the "Hospital Anxiety And Depression (HADS) Scale"
Diagnostic Test: Symptoms - mMRC — Assessment of symptoms by the "modified Medical Research Council (mMRC) scale"
  Groups: Patients with ILD
Diagnostic Test: Sleep quality — Assessment of sleep by the "Pitsburg Sleep Quality Index (PSQI)"
Diagnostic Test: Sleepiness — Assessment of sleepiness by the "Epworth Sleepiness Scale"
Diagnostic Test: Inflammatory markers and oxidative stress — blood assessment of inflammatory markers: IL-2, IL-10, IL-6, IL-4 e IL-17A, TNF, Interferon-γ, CK and CRP.
  Blood assessment of oxidative stress: TRAP, SH, SOD, CAT, PON 1, Gpx, MDA, NOx, FOX and AOPP.
Diagnostic Test: Functional performance tests — Timed-up-and-go at usual pace (TUGu) and at a fast pace (TUGf), four-metre gait speed test (4MGS), sit-to-stand test using three protocols: 30 seconds (30sec-STS), one minute (1min-STS) and five-repetition (5rep-STS) and Short Physical Performance Balance (SPPB).

SUMMARY:
This prospective cohort study will investigate whether progression of the interstitial lung diseases is related to specific clinical endpoints and their changes over time. Longitudinal data of patients will be compared to an age-matched control group during a follow-up of at least two years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with interstitial lung disease:

   * Age between 40 and 75 years old upon inclusion;
   * Diagnosis of interstitial lung disease;
   * Clinical stability for at least 4 weeks prior to inclusion;
   * Absence of any comorbidity that interferes with the performance of tests;
2. Age-matched control group:

   * Age between 40 and 75 years old upon inclusion;
   * Absence of any comorbidity that interferes with the performance of tests;

Exclusion Criteria (both groups):

* Participants that present severe or unstable cardiac disease identified during the cardiopulmonary exercise testing;
* Participants with cognitive deficit that interfere with any of the tests;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A non-probabilistic sample (invitation to volunteer) including participants from the urban region of Londrina, Brazil and surroundings.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes of daily steps over time | from date of inclusion until the date of study completion or until the documented date of death from any cause, whichever came first, up to 48 months
  Changes in daily steps (measured using an activity monitor) at every 6-month interval until study completion or end of participation in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Camillo, PT, PhD, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- Universidade Estadual de Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No
The data collected may be used in other studies upon participants' written consent. However, it is not the intention of investigators to share the data publically (In exception of final results of the study after completion)

REFERENCES:
- [Derived] Garcia T, Mantoani LC, Silva H, Zamboti CL, Ribeiro M, Ramos EMC, Pitta F, Camillo CA. Characteristics of Skeletal Muscle Strength in Subjects With Interstitial Lung Disease. Arch Phys Med Rehabil. 2024 Jun;105(6):1099-1105. doi: 10.1016/j.apmr.2024.01.006. Epub 2024 Jan 24. PMID 38272247